CLINICAL TRIAL: NCT06640933
Title: A Phase 1, Randomized, Open-Label, Single-Dose, 6-Period Crossover Study to Evaluate the Pharmacokinetics of BIIB091 Formulations and the Effect of Food in Healthy Participants
Brief Title: A Study to Find Out How Different Forms of BIIB091 is Processed in The Body With and Without Food in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 257HV106
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — BIIB091

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- BIIB091 IR (Experimental): Participants will receive BIIB091 IR tablets on Day 1 of its respective period, with food.
  Interventions: Drug: BIIB091
- BIIB091 GR-slow (Experimental): Participants will receive BIIB091 GR-slow tablets on Day 1 of its respective period, with food.
  Interventions: Drug: BIIB091
- BIIB091 GR-fast (Experimental): Participants will receive BIIB091 GR-fast tablets on Day 1 of its respective period, with food.
  Interventions: Drug: BIIB091
- BIIB091 ER-slow (Experimental): Participants will receive BIIB091 ER-slow tablets on Day 1 of its respective period, with food.
  Interventions: Drug: BIIB091
- BIIB091 ER-fast (Experimental): Participants will receive BIIB091 ER-fast tablets on Day 1 of its respective period, with food.
  Interventions: Drug: BIIB091
- BIIB091 ER-slow Fasted (Experimental): Participants will receive BIIB091 ER-slow tablets on Day 1 of its respective period, without food.
  Interventions: Drug: BIIB091

INTERVENTIONS:
Drug: BIIB091 — Administered as specified in the treatment arm.

SUMMARY:
In this study, researchers will learn how the body processes new tablet forms of BIIB091 when taken with and without food. One new form of BIIB091 is an "extended release" tablet, also known as "ER." This form helps release BIIB091 slowly and consistently, helping to keep steady drug levels in the body for longer. The other new form is a "gastro-retentive" tablet, also known as "GR." This form has a special coating that swells and allows BIIB091 to stay in the stomach longer. For both GR and ER tablets, there are also "slow" and "fast" forms that change how quickly BIIB091 is released into the body. But, eating food with these tablets may affect how much BIIB091 is in the body.

The main objective of this study is to learn how 2 new forms of BIIB091, which are released into the body at different rates, are processed in the body. Researchers also want to learn how these new forms compare to the "immediate release" tablet, also known as "IR". This form delivers BIIB091 immediately into the body.

The main question researchers want to answer in this study is:

* How does the body process different tablet forms of BIIB091 with or without food?

Researchers will also learn more about:

* How the body processes the 2 new tablet forms of BIIB091 with food compared to the IR tablet form with food
* How the body processes the ER tablet form of BIIB091 with food compared to without food
* Any medical problems the participants have during the study
* Any changes in the participants' overall health during the study

This study will be done as follows:

* Participants will be screened to check if they can join the study. The screening period will be up to 22 days, after which eligible participants will check into their study research center.
* Participants will be randomly assigned to 1 of 6 groups. In each group, the participants will take the below tablet forms, but in different orders:

  * Immediate-Release (IR)
  * Gastro-Retentive slow (GR-slow)
  * Gastro-Retentive fast (GR-fast)
  * Extended-Release slow (ER-slow)
  * Extended-Release fast (ER-fast)
  * ER-slow, without food
* Each period includes the participant taking a single dose of what they were assigned to on the first day. There will be 3 days of no dosing in each period. The participant will then move to the next tablet form assigned. This will continue until each participant has taken a single dose of each of the 6 tablet forms.
* Participants will remain at their study research center for 25 days for the treatment periods. Afterwards, there will be follow-up visit 11 to 14 days after each participant's last dose. Each participant will be in the study for up to 57 days.

DETAILED DESCRIPTION:
The primary objective of this study is to characterize the pharmacokinetics (PK) of BIIB091 after a single oral dose of different BIIB091 formulations with or without food conditions in healthy participants.

The secondary objectives of this study are: to compare the exposure of BIIB091 after a single oral dose of 4 new BIIB091 formulations (GR-fast, GR-slow, ER-fast, ER-slow) with a moderate-fat meal versus a single oral dose of BIIB091 IR tablets with a moderate-fat meal in healthy participants; to compare the exposure of BIIB091 after a single oral dose of BIIB091 ER-slow formulation with a moderate-fat meal versus under fasting conditions in healthy participants; to evaluate the safety and tolerability of BIIB091 after a single oral dose of different BIIB091 formulations with or without food conditions in healthy participants.

ELIGIBILITY:
Key Inclusion Criteria:

* Have a body mass index (BMI) of 18 to 32 kilograms per meter square (kg/m^2), inclusive, and a total body weight >50 kg, Screening and Day -1.
* Negative polymerase chain reaction (PCR) test result for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) at Check-in (Day -1).
* For Japanese participants:

  * Have biological parents and grandparents of Japanese origin.
  * If living outside of Japan for more than 5 years, must not have significantly modified diet since leaving Japan.

Key Exclusion Criteria:

* History of any clinically significant cardiac, endocrine,gastrointestinal (GI), hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, or renal disease or other major disease, as determined by the Investigator.
* History of torsades de pointes or additional risk factors for torsades de pointes.
* Chronic, recurrent, or serious infection (e.g., pneumonia, septicemia), as determined by the Investigator, within 90 days prior to Screening or between Screening and Day -1.

NOTE: Other protocol-defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2024-10-16 (Actual); Primary Completion 2025-02-07 (Actual); Study Completion 2025-02-07 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve From Time Zero to Time of the Last Measurable Concentration (AUClast) of BIIB091 | Predose and at multiple timepoints postdose (up to Day 4)
AUC from Time Zero to Infinity (AUCinf) of BIIB091 | Predose and at multiple timepoints postdose (up to Day 4)
Maximum Observed Concentration (Cmax) of BIIB091 | Predose and at multiple timepoints postdose (up to Day 4)
Time to Reach Cmax (Tmax) of BIIB091 | Predose and at multiple timepoints postdose (up to Day 4)
Elimination Half-Life (t½) of BIIB091 | Predose and at multiple timepoints postdose (up to Day 4)
Time of Last Measurable Concentration (Tlast) of BIIB091 | Predose and at multiple timepoints postdose (up to Day 4)
Concentration of BIIB091 at 12 hours Postdose (C12h) | At multiple timepoints postdose (up to 12 hours)
Apparent Clearance (CL/F) of BIIB091 | Predose and at multiple timepoints postdose (up to Day 4)
Apparent Volume of Distribution During the Terminal Elimination (VZ/F) of BIIB091 | Predose and at multiple timepoints postdose (up to Day 4)

SECONDARY OUTCOMES:
Geometric Mean Ratio (GMR) of AUClast of BIIB091 | Predose and at multiple timepoints postdose (up to Day 4)
GMR of AUCinf of BIIB091 | Predose and at multiple timepoints postdose (up to Day 4)
GMR of Cmax of BIIB091 | Predose and at multiple timepoints postdose (up to Day 4)
GMR of C12h of BIIB091 | At multiple timepoints postdose (up to 12 hours)
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day 1 up to end of study follow-up (up to 35 days)
Number of Participants With Clinically Significant Vital Signs Abnormalities | From Day 1 up to end of study follow-up (up to 35 days)
Number of Participants With Electrocardiogram (ECG) Abnormalities | From Day 1 up to Day 4
Number of Participants With Clinically Significant Laboratory Assessment Abnormalities | At Days 4, 25 and during follow-up (up to 35 days)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (2):
- United States (2):
  - PPD Las Vegas Research Unit, Las Vegas, Nevada
  - PPD Clinical Research Unit, Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/